CLINICAL TRIAL: NCT02625597
Title: An In Vivo Assessment of the Effects of Using Different Implant Abutment Occluding Materials on Implant Microleakage and the Peri-Implant Microbiome
Brief Title: Assessment of the Effects of Different Implant Abutment Occluding Materials on Dental Implant Health Parameters and Microbiology
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stony Brook University (Other)
Responsible Party: Principal Investigator, Julio Carrion, Assistant Professor, Stony Brook University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 409069
Record Dates: First submitted 2015-11-29; First posted 2015-12-09 (Estimated); Last update posted 2015-12-09 (Estimated); Status verified 2015-12

CONDITIONS: Peri-Implantitis; Dental Implant Failed; Dental Implant Failure Nos
MeSH Terms: conditions — Peri-Implantitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dental Materials (Experimental)
  Interventions: Device: Cotton Pellet; Device: Polytetrafluoroethylene Tape; Device: Synthetic Foam; Device: Polyvinylsiloxane

INTERVENTIONS:
Device: Cotton Pellet
  Other Names: Richmond Dental Bleached Cotton
Device: Polytetrafluoroethylene Tape
  Other Names: Teflon; Merco M55 Thread Seal Tape
Device: Synthetic Foam
  Other Names: Jordco Endoring Foam Inserts
Device: Polyvinylsiloxane
  Other Names: Dentsply Aquasil

SUMMARY:
The primary purpose of this study is to determine what effect, if any, do different dental materials used to seal the prosthetic screw channels of implant supported restorations have on dental implant health parameters and microbiology.

ELIGIBILITY:
Inclusion Criteria:

* Fully edentulous patient
* Patient has at least one arch restored with a full-arch dental supported prosthesis

Exclusion Criteria:

* poor oral hygiene and motivation (as determined with prosthesis in place)
* uncontrolled diabetes
* pregnant or lactating
* substance abusers
* current smokers
* psychiatric problems or unrealistic expectations
* acute infection in the area intended for implant sealing
* positive to HIV and hepatitis B and C
* affected by autoimmune diseases
* under chronic treatment with steroids or non-steroidal anti-inflammatory drugs.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2013-11; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
Probing Depth | 6 months

SECONDARY OUTCOMES:
Gingival Index | 6 Months
Plaque Index | 6 Months
Microbial DNA Composition of the Peri-Implant Sulcus Assessed By PCR and Sequencing Protocols | 6 Months
Microbial DNA Composition on the Dental Materials Assessed By PCR and Sequencing Protocols | 6 Months

CONTACTS AND LOCATIONS:
Overall Officials: Julio A Carrion, DMD, PhD, Principal Investigator — Stony Brook University
Locations (1):
- School of Dental Medicine of Stony Brook University, Stony Brook, New York, United States

REFERENCES:
- [Background] Tarica DY, Alvarado VM, Truong ST. Survey of United States dental schools on cementation protocols for implant crown restorations. J Prosthet Dent. 2010 Feb;103(2):68-79. doi: 10.1016/S0022-3913(10)00016-8. PMID 20141811
- [Background] Moraguez OD, Belser UC. The use of polytetrafluoroethylene tape for the management of screw access channels in implant-supported prostheses. J Prosthet Dent. 2010 Mar;103(3):189-91. doi: 10.1016/S0022-3913(10)60029-7. PMID 20188242
- [Background] Peri-implant mucositis and peri-implantitis: a current understanding of their diagnoses and clinical implications. J Periodontol. 2013 Apr;84(4):436-43. doi: 10.1902/jop.2013.134001. No abstract available. PMID 23537178
- [Background] Froum SJ, Rosen PS. A proposed classification for peri-implantitis. Int J Periodontics Restorative Dent. 2012 Oct;32(5):533-40. PMID 22754901
- [Background] Zitzmann NU, Berglundh T. Definition and prevalence of peri-implant diseases. J Clin Periodontol. 2008 Sep;35(8 Suppl):286-91. doi: 10.1111/j.1600-051X.2008.01274.x. PMID 18724856
- [Background] Atieh MA, Alsabeeha NH, Faggion CM Jr, Duncan WJ. The frequency of peri-implant diseases: a systematic review and meta-analysis. J Periodontol. 2013 Nov;84(11):1586-98. doi: 10.1902/jop.2012.120592. Epub 2012 Dec 13. PMID 23237585
- [Background] Daubert DM, Weinstein BF, Bordin S, Leroux BG, Flemming TF. Prevalence and predictive factors for peri-implant disease and implant failure: a cross-sectional analysis. J Periodontol. 2015 Mar;86(3):337-47. doi: 10.1902/jop.2014.140438. Epub 2014 Nov 21. PMID 25415249
- [Background] Tomasi C, Derks J. Clinical research of peri-implant diseases--quality of reporting, case definitions and methods to study incidence, prevalence and risk factors of peri-implant diseases. J Clin Periodontol. 2012 Feb;39 Suppl 12:207-23. doi: 10.1111/j.1600-051X.2011.01831.x. PMID 22533958
- [Background] Mombelli A, Decaillet F. The characteristics of biofilms in peri-implant disease. J Clin Periodontol. 2011 Mar;38 Suppl 11:203-13. doi: 10.1111/j.1600-051X.2010.01666.x. PMID 21323716
- [Background] Mombelli A, Buser D, Lang NP. Colonization of osseointegrated titanium implants in edentulous patients. Early results. Oral Microbiol Immunol. 1988 Sep;3(3):113-20. doi: 10.1111/j.1399-302x.1988.tb00095.x. No abstract available. PMID 3269993
- [Background] Mombelli A, Mericske-Stern R. Microbiological features of stable osseointegrated implants used as abutments for overdentures. Clin Oral Implants Res. 1990 Dec;1(1):1-7. doi: 10.1034/j.1600-0501.1990.010101.x. PMID 2099207
- [Background] Adell R, Lekholm U, Rockler B, Branemark PI, Lindhe J, Eriksson B, Sbordone L. Marginal tissue reactions at osseointegrated titanium fixtures (I). A 3-year longitudinal prospective study. Int J Oral Maxillofac Surg. 1986 Feb;15(1):39-52. doi: 10.1016/s0300-9785(86)80010-2. PMID 3083005
- [Background] Shibli JA, Melo L, Ferrari DS, Figueiredo LC, Faveri M, Feres M. Composition of supra- and subgingival biofilm of subjects with healthy and diseased implants. Clin Oral Implants Res. 2008 Oct;19(10):975-82. doi: 10.1111/j.1600-0501.2008.01566.x. PMID 18828812
- [Background] Kumar PS, Mason MR, Brooker MR, O'Brien K. Pyrosequencing reveals unique microbial signatures associated with healthy and failing dental implants. J Clin Periodontol. 2012 May;39(5):425-33. doi: 10.1111/j.1600-051X.2012.01856.x. Epub 2012 Mar 14. PMID 22417294
- [Background] Danser MM, van Winkelhoff AJ, van der Velden U. Periodontal bacteria colonizing oral mucous membranes in edentulous patients wearing dental implants. J Periodontol. 1997 Mar;68(3):209-16. doi: 10.1902/jop.1997.68.3.209. PMID 9100195
- [Background] Sachdeo A, Haffajee AD, Socransky SS. Biofilms in the edentulous oral cavity. J Prosthodont. 2008 Jul;17(5):348-56. doi: 10.1111/j.1532-849X.2008.00301.x. PMID 18355168
- [Background] Mombelli A, Marxer M, Gaberthuel T, Grunder U, Lang NP. The microbiota of osseointegrated implants in patients with a history of periodontal disease. J Clin Periodontol. 1995 Feb;22(2):124-30. doi: 10.1111/j.1600-051x.1995.tb00123.x. PMID 7775668
- [Background] Pontoriero R, Tonelli MP, Carnevale G, Mombelli A, Nyman SR, Lang NP. Experimentally induced peri-implant mucositis. A clinical study in humans. Clin Oral Implants Res. 1994 Dec;5(4):254-9. doi: 10.1034/j.1600-0501.1994.050409.x. PMID 7640340
- [Background] Mombelli A, van Oosten MA, Schurch E Jr, Land NP. The microbiota associated with successful or failing osseointegrated titanium implants. Oral Microbiol Immunol. 1987 Dec;2(4):145-51. doi: 10.1111/j.1399-302x.1987.tb00298.x. No abstract available. PMID 3507627
- [Background] Rutar A, Lang NP, Buser D, Burgin W, Mombelli A. Retrospective assessment of clinical and microbiological factors affecting periimplant tissue conditions. Clin Oral Implants Res. 2001 Jun;12(3):189-95. doi: 10.1034/j.1600-0501.2001.012003189.x. PMID 11359474
- [Background] Salcetti JM, Moriarty JD, Cooper LF, Smith FW, Collins JG, Socransky SS, Offenbacher S. The clinical, microbial, and host response characteristics of the failing implant. Int J Oral Maxillofac Implants. 1997 Jan-Feb;12(1):32-42. PMID 9048452
- [Background] Persson GR, Renvert S. Cluster of bacteria associated with peri-implantitis. Clin Implant Dent Relat Res. 2014 Dec;16(6):783-93. doi: 10.1111/cid.12052. Epub 2013 Mar 25. PMID 23527870
- [Background] Albertini M, Lopez-Cerero L, O'Sullivan MG, Chereguini CF, Ballesta S, Rios V, Herrero-Climent M, Bullon P. Assessment of periodontal and opportunistic flora in patients with peri-implantitis. Clin Oral Implants Res. 2015 Aug;26(8):937-941. doi: 10.1111/clr.12387. Epub 2014 Apr 10. PMID 24720498
- [Background] Salvi GE, Aglietta M, Eick S, Sculean A, Lang NP, Ramseier CA. Reversibility of experimental peri-implant mucositis compared with experimental gingivitis in humans. Clin Oral Implants Res. 2012 Feb;23(2):182-190. doi: 10.1111/j.1600-0501.2011.02220.x. Epub 2011 Aug 2. PMID 21806683
- [Background] Lindhe J, Meyle J; Group D of European Workshop on Periodontology. Peri-implant diseases: Consensus Report of the Sixth European Workshop on Periodontology. J Clin Periodontol. 2008 Sep;35(8 Suppl):282-5. doi: 10.1111/j.1600-051X.2008.01283.x. PMID 18724855
- [Background] Charalampakis G, Leonhardt A, Rabe P, Dahlen G. Clinical and microbiological characteristics of peri-implantitis cases: a retrospective multicentre study. Clin Oral Implants Res. 2012 Sep;23(9):1045-54. doi: 10.1111/j.1600-0501.2011.02258.x. Epub 2011 Aug 3. PMID 22092339
- [Background] Quirynen M, van Steenberghe D. Bacterial colonization of the internal part of two-stage implants. An in vivo study. Clin Oral Implants Res. 1993 Sep;4(3):158-61. doi: 10.1034/j.1600-0501.1993.040307.x. PMID 8297964
- [Background] Passos SP, Gressler May L, Faria R, Ozcan M, Bottino MA. Implant-abutment gap versus microbial colonization: Clinical significance based on a literature review. J Biomed Mater Res B Appl Biomater. 2013 Oct;101(7):1321-8. doi: 10.1002/jbm.b.32945. Epub 2013 May 10. PMID 23661560
- [Background] Persson LG, Lekholm U, Leonhardt A, Dahlen G, Lindhe J. Bacterial colonization on internal surfaces of Branemark system implant components. Clin Oral Implants Res. 1996 Jun;7(2):90-5. doi: 10.1034/j.1600-0501.1996.070201.x. PMID 9002826
- [Background] Nascimento Cd, Ikeda LN, Pita MS, Pedroso e Silva RC, Pedrazzi V, Albuquerque RF, Ribeiro RF. Marginal fit and microbial leakage along the implant-abutment interface of fixed partial prostheses: An in vitro analysis using Checkerboard DNA-DNA hybridization. J Prosthet Dent. 2015 Dec;114(6):831-8. doi: 10.1016/j.prosdent.2015.05.009. Epub 2015 Sep 8. PMID 26359546
- [Background] Gross M, Abramovich I, Weiss EI. Microleakage at the abutment-implant interface of osseointegrated implants: a comparative study. Int J Oral Maxillofac Implants. 1999 Jan-Feb;14(1):94-100. PMID 10074758
- [Background] Ericsson I, Persson LG, Berglundh T, Marinello CP, Lindhe J, Klinge B. Different types of inflammatory reactions in peri-implant soft tissues. J Clin Periodontol. 1995 Mar;22(3):255-61. doi: 10.1111/j.1600-051x.1995.tb00143.x. PMID 7790533
- [Background] Broggini N, McManus LM, Hermann JS, Medina R, Schenk RK, Buser D, Cochran DL. Peri-implant inflammation defined by the implant-abutment interface. J Dent Res. 2006 May;85(5):473-8. doi: 10.1177/154405910608500515. PMID 16632764
- [Background] Covani U, Marconcini S, Crespi R, Barone A. Bacterial plaque colonization around dental implant surfaces. Implant Dent. 2006 Sep;15(3):298-304. doi: 10.1097/01.id.0000226823.58425.19. PMID 16966904
- [Background] da Silva-Neto JP, Nobilo MA, Penatti MP, Simamoto PC Jr, das Neves FD. Influence of methodologic aspects on the results of implant-abutment interface microleakage tests: a critical review of in vitro studies. Int J Oral Maxillofac Implants. 2012 Jul-Aug;27(4):793-800. PMID 22848880
- [Background] Taylor RC, Ghoneim AS, McGlumphy EA. An esthetic technique to fill screw-retained fixed prostheses. J Oral Implantol. 2004;30(6):384-5. doi: 10.1563/0681.1. PMID 15641458
- [Background] Park SD, Lee Y, Kim YL, Yu SH, Bae JM, Cho HW. Microleakage of different sealing materials in access holes of internal connection implant systems. J Prosthet Dent. 2012 Sep;108(3):173-80. doi: 10.1016/S0022-3913(12)60143-7. PMID 22944313
- [Background] Klindworth A, Pruesse E, Schweer T, Peplies J, Quast C, Horn M, Glockner FO. Evaluation of general 16S ribosomal RNA gene PCR primers for classical and next-generation sequencing-based diversity studies. Nucleic Acids Res. 2013 Jan 7;41(1):e1. doi: 10.1093/nar/gks808. Epub 2012 Aug 28. PMID 22933715
- [Background] Socransky SS, Haffajee AD. Periodontal microbial ecology. Periodontol 2000. 2005;38:135-87. doi: 10.1111/j.1600-0757.2005.00107.x. No abstract available. PMID 15853940
- [Background] da Silva ES, Feres M, Figueiredo LC, Shibli JA, Ramiro FS, Faveri M. Microbiological diversity of peri-implantitis biofilm by Sanger sequencing. Clin Oral Implants Res. 2014 Oct;25(10):1192-9. doi: 10.1111/clr.12231. Epub 2013 Jul 12. PMID 23845046